CLINICAL TRIAL: NCT00500305
Title: The Use of B-type Natriuretic Peptide (BNP) to Predict Closure of a Patent Ductus Arteriosus (PDA) in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10946
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Indomethacin Therapy; Patent Ductus Arteriosus
Keywords: indomethacin therapy; patent ductus arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Withhold standard INDO dose if BNP < 100 pg/ml

SUMMARY:
A patent ductus arteriosus (PDA) is associated with increased morbidity in premature infants. Standard indomethacin treatment is associated with intestinal and renal morbidity. B-type natriuretic peptide is elevated in significant PDAs. This study will determine whether BNP guided therapy could reduce doses of indomethacin.

ELIGIBILITY:
Inclusion Criteria:

* Infants with echocardiographically confirmed PDA
* Infants determined by attending physician to require PDA closure

Exclusion Criteria:

* infants with congenital hearts disease
* infants with creatinine value > 2.0

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2004-04; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Number of indomethacin doses given on study | 2 days

SECONDARY OUTCOMES:
rate of PDA ligation | Discharge from NICU
Rate of Chronic lung disease | 36 weeks corrected gestational age

CONTACTS AND LOCATIONS:
Overall Officials: D Sc Lim, MD, Principal Investigator — University of Virginia